CLINICAL TRIAL: NCT05146206
Title: Patient Satisfaction and Sensory Attributes of Nasal Spray Treatments for Allergic Rhinitis
Brief Title: Patient Satisfaction and Sensory Attributes Allergic Rhinitis Nasal Spray
Status: Completed | Type: Observational
Sponsor: Community and Patient Preference Research Pty Ltd (Industry)
Collaborators: Seqirus (Industry); Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20210902_2
Record Dates: First submitted 2021-11-10; First posted 2021-12-06 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Allergic Rhinitis
Keywords: Patient preference; Best-Worst Scaling; Treatment attributes
MeSH Terms: conditions — Rhinitis, Allergic; Patient Preference | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients on RYALTRIS: Patients who are currently using RYALTRIS nasal spray.
  Interventions: Other: Observational
- Patients on DYMISTA: Patients who are currently using DYMISTA nasal spray.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — In this observational study, participants initated on RYALTRIS/DYMISTA nasal spray will complete a cross-sectional online survey that includes a Best-Worst Scaling task to capture their satisfaction and importance of various treatment attributes.

SUMMARY:
The study seeks to understand patients' satisfaction and importance of treatment attributes for Allergic Rhinitis nasal sprays from two brands (RYALTRIS® vs. DYMISTA®).

DETAILED DESCRIPTION:
The study seeks to understand patients' satisfaction and importance of treatment attributes for Allergic Rhinitis nasal sprays from two brands (RYALTRIS® vs. DYMISTA®).

To directly compare patient satisfaction with 2 different Allergic Rhinitis nasal sprays, an observational, cross-sectional study design with 2 independent samples was chosen. Participants will complete an online survey involving a Best-Worst scaling (BWS) task to determine satisfaction and importance index for sensory attributes.

The suggested treatment attributes are informed by a range of previous studies, including those conducted by Meltzer et al 2005 and Price et al 2020, and methodology from CaPPRe's own work in developing indices for importance and satisfaction of treatment attributes using BWS.

ELIGIBILITY:
Inclusion Criteria:

Allergic Rhinitis patients (moderate-to-severe Seasonal Allergic Rhinitis or Perennial Allergic Rhinitis) with or without conjunctivitis who meet the following criteria will be offered the opportunity to participate in the study:

* Patients above 18 years old
* Fluent in English
* Patients initiated on RYALTRIS® or DYMISTA® nasal spray in the last 12 months and currently using treatment
* Willing and able to provide consent to participate

Exclusion Criteria:

* Have reported a loss of taste and/or smell related to COVID-19 (or other medical condition)
* Are employed by a pharmaceutical company (to avoid conflict of interest)
* Are employed by a vaccine company (to avoid conflict of interest)
* Do not have access to the internet (to ensure validity of the data)
* Are unable to read and understand English (to ensure validity of the data)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The primary population will be patients with moderate to severe SAR or PAR with or without conjunctivitis in Australia who have been initiated on RYALTRIS® or DYMISTA® in that last 12 months.
  The expected sample size is between 200 to 400 patients. 100-200 patients initiated on RYALTRIS® and 100-200 patients initiated on DYMISTA® nasal spray in the last 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Fifer, PhD, Principal Investigator — Community and Patient Preference Research Pty Ltd
Locations (1):
- Community and Patient Preference Research Pty Ltd, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Australian Institute of Health and Welfare 2019. Allergic rhinitis ('hay fever'). Cat. no. PHE 257. Canberra: AIHW. Viewed 01 May 2020, https://www.aihw.gov.au/reports/chronic-respiratory-conditions/allergic-rhinitis-hay-fever/contents/allergic-rhinitis
- [Background] Meltzer EO, Bardelas J, Goldsobel A, Kaiser H. A preference evaluation study comparing the sensory attributes of mometasone furoate and fluticasone propionate nasal sprays by patients with allergic rhinitis. Treat Respir Med. 2005;4(4):289-96. doi: 10.2165/00151829-200504040-00007. PMID 16086602
- [Background] Meltzer EO, Garadi R, Laforce C, Chadwick SJ, Berger WE, Gross G, Edwards MR, Crenshaw K, Wall GM. Comparative study of sensory attributes of two antihistamine nasal sprays: olopatadine 0.6% and azelastine 0.1%. Allergy Asthma Proc. 2008 Nov-Dec;29(6):659-68. doi: 10.2500/aap.2008.29.3181. Epub 2008 Dec 6. PMID 19144261
- [Background] Meltzer EO, Hadley J, Blaiss M, Benninger M, Kimel M, Kleinman L, Dupclay L, Garcia J, Leahy M, Georges G. Development of questionnaires to measure patient preferences for intranasal corticosteroids in patients with allergic rhinitis. Otolaryngol Head Neck Surg. 2005 Feb;132(2):197-207. doi: 10.1016/j.otohns.2004.10.010. PMID 15692526
- [Background] Price D, Klimek L, Galffy G, Emmeluth M, Koltun A, Kopietz F, Nguyen DT, van Weissenbruch R, Pohl W, Kuhl HC, Scadding G, Mullol J. Allergic rhinitis and asthma symptoms in a real-life study of MP-AzeFlu to treat multimorbid allergic rhinitis and asthma. Clin Mol Allergy. 2020 Aug 6;18:15. doi: 10.1186/s12948-020-00130-9. eCollection 2020. PMID 32782442
- [Background] Louviere, J., Flynn, T., Marley, A., 2015. References. In Best-Worst Scaling: Theory, Methods and Applications Cambridge University, Cambridge, pp. 316-331
- [Background] Muhlbacher AC, Kaczynski A, Zweifel P, Johnson FR. Experimental measurement of preferences in health and healthcare using best-worst scaling: an overview. Health Econ Rev. 2016 Dec;6(1):2. doi: 10.1186/s13561-015-0079-x. Epub 2016 Jan 8. PMID 26743636

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As some eligible participants did not complete the online survey, more participants had to be recruited to meet the target sample size. This was done to ensure there was enough statistical power for analyses.
Period: Overall Study
Arm/Group | Patients on RYALTRIS | Patients on DYMISTA
Started | 98 | 328
Completed | 98 | 328
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: As this was a non-interventional study, all participants were already initiated on their treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients on RYALTRIS | Patients on DYMISTA | Total
Number analyzed (Participants) | 98 | 328 | 426
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 292 | 384
  >=65 years | 6 | 36 | 42
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 44 | 249 | 293
  Gender: Male | 54 | 77 | 131
  Gender: Non-binary/gender fluid | 0 | 1 | 1
  Gender: Prefer not to answer | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Treatment Satisfaction Index [Mean (Standard Deviation); unit: units on a scale ranging from 0 to 100.] — The Treatment Satisfaction Index measures overall satisfaction with the current treatment. The scale ranges from 0 to 100. Higher values represent greater overall satisfaction with the current treatment.
  units on a scale ranging from 0 to 100. | 68.26 (13.76) | 62.78 (12.60) | 64.04 (13.07)

OUTCOME MEASURES:

1. Primary Outcome: Overall Best-Worst Scaling Task Index Score (Treatment Satisfaction Index Score)
Description: The primary study endpoint is the overall index score from the Best Worst Scaling exercise, to reflect satisfaction and importance of treatment attributes of the RYALTRIS® and DYMISTA® nasal spray.
  Index scores from the Best Worst Scaling exercise range from 0 to 100, with higher scores indicating higher satisfaction of treatment attributes.
Time Frame: Cross-sectional - through study completion, an average of 3 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Participants Using Ryaltris (OLO/MOM): Participants using Ryaltris (OLO/MOM)
- Participants Using Dymista (AZE/FLU): Participants using Dymista (AZE/FLU)
Arm/Group | Participants Using Ryaltris (OLO/MOM) | Participants Using Dymista (AZE/FLU)
Number analyzed (Participants) | 98 | 328
units on a scale | 68.26 (1.39) | 62.78 (0.70)
Statistical Analysis 1: Comparison: Participants Using Ryaltris (OLO/MOM) vs Participants Using Dymista (AZE/FLU); Test type: Other; p < .001, ANOVA

2. Secondary Outcome: Rescaled Scores From Best-Worst Scaling Task
Description: Secondary study endpoints were the rescaled Best Worst Scaling domain scores from the Best Worst Scaling exercise (i.e., scores for each of the domains on satisfaction and importance).
  Rescaled Best-Worst Scaling domain scores range from 0 to 10 and represent the satisfaction and importance of each domain. Higher satisfaction rescaled scores indicate higher satisfaction on a treatment attribute. Higher importance rescaled scores indicate higher importance of the treatment attribute. Higher rescaled satisfaction and importance scores suggest a better outcome since participants are satisfied and more likely to adhere to their current treatment.
Time Frame: Cross-sectional - through study completion, an average of 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Participants Using Ryaltris (OLO/MOM) | Participants Using Dymista (AZE/FLU)
Number analyzed (Participants) | 98 | 328
units on a scale
  Satisfaction - Immediate taste of medication | 6.12 (0.62) | 4.66 (0.26)
  Satisfaction - Aftertaste of medication | 5.84 (0.59) | 4.21 (0.23)
  Satisfaction - Smell of medication | 6.31 (0.64) | 5.55 (0.31)
  Satisfaction - Irritation to your nose | 6.05 (0.61) | 5.37 (0.30)
  Satisfaction - Urge to sneeze | 6.35 (0.64) | 5.52 (0.30)
  Satisfaction - Dripping out your nose/down your throat | 6.20 (0.63) | 4.89 (0.27)
  Satisfaction - Dryness of your nose or throat | 6.41 (0.65) | 5.64 (0.31)
  Satisfaction - Convenience (how easy it is to administer) | 7.31 (0.74) | 7.15 (0.39)
  Satisfaction - Fast acting (how quickly it works | 7.55 (0.76) | 7.16 (0.40)
  Satisfaction - Duration of effect (long lasting) | 7.30 (0.74) | 6.89 (0.38)
  Satisfaction - Perceived allergic rhinitis symptom control | 7.38 (0.75) | 7.96 (0.44)
  Importance - Immediate taste of medication | 5.84 (0.59) | 4.63 (0.26)
  Importance - Aftertaste of medication | 5.59 (0.56) | 4.80 (0.27)
  Importance - Smell of medication | 5.20 (0.53) | 3.41 (0.19)
  Importance - Irritation to your nose | 6.08 (0.61) | 5.51 (0.30)
  Importance - Urge to sneeze | 5.88 (0.59) | 4.69 (0.26)
  Importance - Dripping out your nose/down your throat | 6.29 (0.64) | 5.43 (0.30)
  Importance - Dryness of your nose or throat | 6.28 (0.63) | 5.49 (0.30)
  Importance - Convenience (how easy it is to administer) | 6.65 (0.67) | 6.17 (0.34)
  Importance - Fast acting (how quickly it works) | 7.35 (0.74) | 7.48 (0.41)
  Importance - Duration of effect (long lasting) | 7.34 (0.74) | 7.70 (0.43)
  Importance - Perceived allergic rhinitis symptom control | 8.00 (0.81) | 8.86 (0.49)
Statistical Analysis 1: Comparison: Participants Using Ryaltris (OLO/MOM) vs Participants Using Dymista (AZE/FLU); Test type: Other; p < 0.001, MANOVA

ADVERSE EVENTS:
Description: Adverse events data were not collected in this online observational survey as there were no open-text fields.
Arm/Group | Patients on RYALTRIS | Patients on DYMISTA
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT05146206/Prot_SAP_000.pdf